CLINICAL TRIAL: NCT02613351
Title: Leg Muscle Activity and Sensation During Upright Partitioned Exercise Compared to Walking: Propulsion of a 3-wheeled Scooter by Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Muscle Activity and Sensation During Upright Partitioned Leg Exercise in COPD
Acronym: MAPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Directory Respiratory Medicine, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPHC-RG-1Lscoot20151201
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exercise Tolerance; Lung Diseases, Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- scooting (Experimental): incremental test to establish the relationship between leg and breathing heaviness with increasing demand (speed) during scooting
  Interventions: Device: scooting

INTERVENTIONS:
Device: scooting — three-wheeled scooter (Monark 662, Monark Exercise AB Sweden) comprised of a single front wheel that provides steering and two rear wheels that create a wide base of support.

SUMMARY:
The aim of this study is to determine if: the large muscles of the leg, activated during walking, are also active during scooting; whether scooting alters the relationship between leg and breathing heaviness; whether there is evidence of leg fatigue during scooting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD: FEV1 < 80 % and FEV1/FVC < 0.7;
* Able to communicate in English
* Clinically stable

Exclusion Criteria:

* predominant co-morbidities or treatments that might influence the results of exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
slope of the relationship between self-reported breathing and leg heaviness using Borg scale | 1 week
  Borg scale ratings of breathing and leg heaviness will be measured during stepwise incremental speed exercise tests. The relationship between leg and breathing heaviness with increasing demand (speed) is quantified by the slope of the relationship between self-reported breathing and leg heaviness under each condition of customary walking and scooting.

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, MD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- Westpark Health Care Centre, Toronto, Ontario, Canada